CLINICAL TRIAL: NCT04040517
Title: [ASSR] in Hearing Impaired Children With Absent [ABR] Waves
Brief Title: Auditory Steady State Response vsAuditory Brainstem Response
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Galal Ibrahem, resident doctor Alazhar university - Assiut, Assiut University
Other Study IDs: 17100772
Record Dates: First submitted 2019-05-21; First posted 2019-07-31 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Hearing Impaired Children
Keywords: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Evoked potential audiometer — The ASSR [ steady state response] test stimuli are modulated pure tones with insert earphone..
  Other Names: Auditory steady state response

SUMMARY:
All children with hearing loss should have access to resources necessary to reach their maximum potential. The following principles provide the foundation for effective EHDI[Early Hearing Detection & Intervention] systems and have been updated and expanded since the 2000 JCIH [ joint Committee on Infant Hearing ] position statement .

DETAILED DESCRIPTION:
1. All infants should have access to hearing screening using a physiologic measure at no later than 1 month of age.
2. All infants who do not pass the initial hearing screening and the subsequent rescreening should have appropriate audiological and medical evaluations to confirm the presence of hearing loss at no later than 3 months of age.
3. All infants with confirmed permanent hearing loss should receive early intervention services as soon as possible after diagnosis but at no later than 6 months of age. A simplified, single point of entry into an intervention system that is appropriate for children with hearing loss is optimal.

The importance of early identification and habilitation of hearing loss for improved access to auditory stimuli and for positive prognosis of speech and language is well established in the literature . Auditory brain stem response (ABR) is the most commonlly used test in clinical practice to estimate the degree of hearing loss, but the auditory brainstem response (ABR) cannot differentiate between severe and profound SNHL [5], whereas the ASSR can provide threshold information in a frequency-specific manner at intensity levels of 120 dB and higher. This intensity stimulation advantage uniquely qualifies the ASSR for investigation of residual hearing in young and difficult-to-test cochlear implant candidates.

ELIGIBILITY:
Inclusion Criteria:

* Absent ABR [Auditory Breanstem Response] waves .
* normal middle ear function

Exclusion Criteria:

* Ears with otitis media with effusion,
* Preserved otoacuastic emission ,
* Preserved ABR waves .

Ages: 1 Day to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Evaluate of residual hearing function in hearing impaired children with absent ABR waves and normal middle ear pressure.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
A 40 hearing impaired children with absent ABR waves | one year
  evaluation by auditory steady state response (ASSR)

SECONDARY OUTCOMES:
After ASSR evaluation for this patient we can take decision either for hearing aid amplification of for (surgery) cochlear implant . | one year
  evaluation by auditory steady state response (ASSR)

REFERENCES:
- [Background] Wadhera R, Hernot S, Gulati SP, Kalra V. A controlled comparison of auditory steady-state responses and pure-tone audiometry in patients with hearing loss. Ear Nose Throat J. 2017 Oct-Nov;96(10-11):E47-E52. doi: 10.1177/0145561317096010-1109. PMID 29121385